CLINICAL TRIAL: NCT03351374
Title: Web Platform to Integrate Behavioral Health
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Medical Decision Logic, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: N44DA-17-5679
Record Dates: First submitted 2017-11-20; First posted 2017-11-22 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Integrating Behavioral Health
Keywords: behavioral health; software; integration

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Temple Physicians Incorporated: A community-based provider, operating 32 primary care sites
  Interventions: Other: Software
- WhiteBark: For profit entity created by the Indiana Rural Health Association
  Interventions: Other: Software
- Drexel Family Intervention Science: Academic center that developed and deployed Attachment Based Family Therapy (ABFT) assessment, treatment, and prevention models with an interest in adolescents struggling with substance abuse, depression, trauma, and suicidality.
  Interventions: Other: Software
- Bon Secours Health System: A primary care clinic in Baltimore that provides care services to a population in a lower socioeconomic status in downtown Baltimore.
  Interventions: Other: Software
- Howard University Hospital CARES: A project provides free outpatient medical, dental, mental health, nutrition and social services for HIV positive uninsured and underinsured residents of the District of Columbia.
  Interventions: Other: Software

INTERVENTIONS:
Other: Software — multi-module system of web software tools

SUMMARY:
Under this Small Business Innovation Research (SBIR) Phase II project, Research Topic 155, the Contractor will create an integrated multi-module system of web software tools to aid in behavioral health screening, prevention, triage, and tracking in medical, school, and mental health settings.

DETAILED DESCRIPTION:
Health care systems experience problems with lack of tools, lack of knowledge, process variation, and system fragmentation in addressing behavioral health. As an ongoing science-based process for improving care and lowering costs, robust increases in translational capability are needed to re-tool health delivery systems for behavioral health integration. A logic linking translational capability to behavioral health integration as an ongoing shared information process, founded on the core belief that enabling human action with new information technology tools can grow knowledge, is the most powerful way to solve problems and improve health care.

Given these connected and interacting issues and obstacles, the Contractor has developed a solution strategy, building on four tiers of prior innovation and validation:

* The Behavioral Health Screen (BHS);
* BH-Works: the web software delivery of the BHS and new production features from Phase I;
* BH-Works Portal: new production software features from Phase I; and
* BH-Works Services: expertise and professional services to help primary care providers and healthcare systems integrate behavioral health into their organizations and workflows.

ELIGIBILITY:
Inclusion Criteria:

* Potential Mental Health issue

Exclusion Criteria:

* Not Willing to be Screened for mental health issues

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients that enter the health system through primary care clinics, academic medical and behavioral health centers, hospitals, or rural health clinics.
Sampling Method: Non-Probability Sample
Enrollment: 16000 (Estimated)
Dates: Start 2018-09-25 (Estimated); Primary Completion 2019-09-25 (Estimated); Study Completion 2019-09-25 (Estimated)

PRIMARY OUTCOMES:
Increase Provider Integration | 2 Years
  Increase collaboration between Primary Care Physician and mental health series.

SECONDARY OUTCOMES:
Increase Screening | 2 Years
  Increase identification rates of adults with depression and substance abuse problems.
Increase Referrals | 2 Years
  Increase successful referrals to mental health services.

CONTACTS AND LOCATIONS:
Overall Officials: Allen Tien, MD, Principal Investigator — Medical Decision Logic, Inc.
Locations (2):
- United States (2):
  - Fayette Regional, Connersville, Indiana
  - Port Richmond Family Medicine, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No